CLINICAL TRIAL: NCT03597373
Title: Variables Predicting Reintubation After Thymectomy in Patients With Myasthenia Gravis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, GengLong Liu, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: Reintubation
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Myasthenia Gravis
Keywords: Prediction; Myasthenia gravis; Reintubation
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- reintubation: Reestablish of invasive mechanical ventilation
  Interventions: Other: reintubation
- not reintubation: Favourable respiratory function
  Interventions: Other: reintubation

INTERVENTIONS:
Other: reintubation — Reintubation was defied by the reinstitution of invasive mechanical ventilation following extubation at any time

SUMMARY:
Myasthenia gravis (MG) is an autoimmune disease that is characterized by muscle weakness and fatigue. The role of the thymus in MG has been suggested by the evidence that 10% to 15% of patients present with a thymoma and at least 60% with thymus hyperplasia or dysplasia.Beneficial effects of thymectomy in patients with MG have been described in 40% to 90%.Few studies have looked at the incidence of reintubation (not just within 24 hours after extubation), the factors associated with reintubation, and patient outcome.

Premature extubation may lead to hypercarbia, hypoxemia, pulmonary hypertension, right heart failure, and myocardial ischemia. Additionally, it subjects the patient to the physical risks of reintubation, including esophageal intubation, laryngeal trauma, and pulmonary aspiration. The purpose of the present study was to determine the incidence of reintubation, the variables associated with reintubation, and patient outcome

DETAILED DESCRIPTION:
Inclusion was based on the availability of all the following possible predictive pre-operative variables: age, gender, weight, height, body mass index, diabetes, creatinine, duration of MG, severity of MG (based on Osserman's classification), pathological type of MG, history of myasthenic crisis, dose of pyridostigmine, use of a steroid hormone, and use of an immunosuppressant.operative variables: postoperative pulmonary infection, total duration of hospital stay, duration of ICU stay, and duration of postoperative hospital stay. Variables were collected by research assistants and maintained in a computer database.

ELIGIBILITY:
Inclusion Criteria:

* younger than 75 years
* absence of heart failure as the primary indication for mechanical ventilation •Acute Physiology and Chronic Health Evaluation (APACHE) II score less than 12 points on day of extubation
* body mass index less than 30

Exclusion Criteria:

•preoperative moderate-to-severe chronic obstructive pulmonary disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with myasthenia gravis undergoing thymectomy
Sampling Method: Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Risk Factors for Reintubation | an average of 30 days
  the reintubation rate was analyzed with logistic regression

CONTACTS AND LOCATIONS:
Overall Officials: Genglong Liu, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Genglong Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided